CLINICAL TRIAL: NCT05516459
Title: Prospective Monitoring of BNT162b2 Second Vaccination Booster for Prevention of the COVID-19 Infection in Health Care Workers (HCW)
Brief Title: Prospective Monitoring of BNT162b2 Second Vaccination Booster Effects in Health Care Workers (HCW)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Victor Novack, Head of Internal Department H, Soroka University Medical Center
Other Study IDs: SCRC22001
Record Dates: First submitted 2022-08-21; First posted 2022-08-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — * Blood drawn for PBMC and antibody testing:
    * Will be at ONLY at Soroka Medical Center. Subjects who were not part of the PBMC group and are willing to participate, will be asked again to sign inform consent.
    * Subjects participating in this part will have 30 ml (3 vials of 9 ml and 1 vial of 3 ml) of blood drawn for PBMC and antibody testing. Others will have blood draw of three 5 ml vials, for antibody testing.
  * A nasal and mouth swab will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Three doses of vaccination: Subjects received three pfizer BNT162b2 vaccination at least four month before recruitment
- Four doses of vaccination: Subjects received three pfizer BNT162b2 vaccination at least four month before recruitment and decided to receive another dose at time of recruitment or followup
  Interventions: Biological: Pfizer BNT162b2 Vaccine

INTERVENTIONS:
Biological: Pfizer BNT162b2 Vaccine — The Pfizer-BioNTech COVID-19 vaccine (INN: tozinameran), sold under the brand name Comirnaty, is an mRNA-based COVID-19 vaccine developed by the German biotechnology company BioNTech. For its development, BioNTech collaborated with American company Pfizer to carry out clinical trials, logistics, and manufacturing. It is authorized for use in people aged five years and older in some jurisdictions, twelve years and older in some jurisdictions, and for people sixteen years and older in other jurisdictions, to provide protection against COVID-19, caused by infection with the SARS-CoV-2 virus. The vaccine is given by intramuscular injection. It is composed of nucleoside-modified mRNA (modRNA) encoding a mutated form of the full-length spike protein of SARS-CoV-2, which is encapsulated in lipid nanoparticles. Initial advice indicated that vaccination required two doses given 21 days apart, but the interval was later extended to up to 42 days in the US, and up to four months in Canada
  Groups: Four doses of vaccination

SUMMARY:
The SARS-CoV-2 virus causes severe respiratory illness and is an ongoing global pandemic. On December 12, 2020 the FDA approved Pfizer's BioNTech vaccine BNT162b2 which is a messenger RNA type of vaccine for use. This vaccine has shown in numerous studies the ability to induce a strong immune response and provide both humeral and cellular protection against wild type, alpha and delta variants of SARS-CoV2 virus.

In Israel the national vaccine operation began in mid-December 2020 which included 2 initial doses three weeks apart. In August 2021 a first booster (3rd dose) was provided to enhance protection and due to reports of reduced immune response and clinical protection. Several studies have demonstrated that over time there is a decay in the antibody levels, and with them reduced protection.

Recently a new variant of concern has been identified (Omicron) and is causing a surge of infections worldwide. There is lack of knowledge regarding the effectiveness of the current schedule of vaccine against this new variant and whether a second booster (4th dose) will provide higher levels of clinical protection against this variant, currently the ministry of health is considering recommendations for a fourth dose for HCW.

The purpose of this study is to examine whether a fourth dose of vaccination will provide better protection against infection and clinical disease.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. Healthcare worker in one of the Clalit Health Services Medical centers and is at least 18 years of age.
3. Completed three doses of BNT162b2 according to MOH guidelines.
4. Third dose was given at least 4 months prior to enrollment.

Exclusion Criteria:

1. History of COVID-19 infection.
2. History of being treated or is currently being treated for any type of Malignancies or other co-morbid conditions that may result in protocol non-compliance.
3. Currently or in the past three months was treated with any type of Immune suppression medication (including chemotherapy, immunomodulatory drugs, biological agents that affect the immune system, any immunosuppressive drug such as corticosteroids).
4. Received in the past 4 months monoclonal antibodies of any type.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be screened at each participating medical center. The study population will be enrolled according to the following inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of positive PCR test for SARS-COV2 | 30 days
  Percent Positive PCR test
Proportion of positive PCR test for SARS-COV2 | 60 days
  Percent Positive PCR test
Proportion of positive PCR test for SARS-COV2 | 90 days
  Percent Positive PCR test
Proportion of positive PCR test for SARS-COV2 | 120 days
  Percent Positive PCR test
Proportion of positive PCR test for SARS-COV2 | 150 days
  Percent Positive PCR test

SECONDARY OUTCOMES:
Proportion of symptomatic COVID 19 infection | 30 days
  Percent Positive PCR test
Proportion of symptomatic COVID 19 infection | 90 days
  Percent Positive PCR test
Proportion of symptomatic COVID 19 infection | 182 days
  Percent Positive PCR test
Proportion of COVID 19 infection requiring hospitalization | 30days
  Percent Positive PCR test
Proportion of COVID 19 infection requiring hospitalization | 90 days
  Percent Positive PCR test
Proportion of COVID 19 infection requiring hospitalization | 182 days
  Percent Positive PCR test
Levels of binding and neutralizing activity and avidity of the antibodies | 30 days
  binding antibody units per mL
Levels of binding and neutralizing activity and avidity of the antibodies | 60 days
  50 Percent neutralization titer
Levels of binding and neutralizing activity and avidity of the antibodies | 90 days
  50 Percent neutralization titer
Levels of binding and neutralizing activity and avidity of the antibodies | 120 days
  50 Percent neutralization titer
Levels of binding and neutralizing activity and avidity of the antibodies | 150 days
  50 Percent neutralization titer
Levels of binding and neutralizing activity and avidity of the antibodies | 180 days
  50 Percent neutralization titer
Composite endpoint of serious adverse events | 14 days following the booster vaccination
  Percent Positive Anaphylaxis, Myocarditis

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka UMC, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No
Unidentified participant data will be made available when the study is complete upon requests directed to the corresponding author. Proposals will be reviewed and approved by the sponsor, investigator, and collaborators on the basis of scientific merit. After approval of a proposal, data can be shared through a secure online platform after signing a data access agreement. All data will be made available for a minimum of 5 years from the end of the study.

DOCUMENTS (1):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT05516459/Prot_000.pdf